CLINICAL TRIAL: NCT07098793
Title: Cough Monitoring in COPD:a Mixed Methods Observational Study
Brief Title: Cough Monitoring in COPD
Status: Completed | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Other Study IDs: COPD2023
Record Dates: First submitted 2023-09-05; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-03

CONDITIONS: Cough; COPD; COPD Exacerbation
MeSH Terms: conditions — Cough; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with COPD: Patients with frequent exacerbations of COPD
  Interventions: Device: Cough monitoring

INTERVENTIONS:
Device: Cough monitoring — continuous recording of cough in patients sleeping area for 90-180 days

SUMMARY:
This is an observational study designed to learn about symptoms of cough and how changes in cough may be associated with the beginning of a COPD exacerbation (acute worsening of symptoms.

The Investigators are looking to recruit patients diagnosed with COPD who have had two or more exacerbations of their disease within the last year requiring treatment with antibiotics or corticosteroids.

The main question aimed to be answered is whether the cough monitor can detect changes in a patient's clinical condition.

Patients will be screened for participation in the study and a medical history will be taken alongside details of current medications, height, weight, vital signs as well and smoking status.

The patients will be asked to complete 3 questionnaires and the cough monitor will be installed in the room within their home where they sleep.

Patients will be asked to complete a daily diary for 90 to a maximum of 180 days and leave the monitor recording cough throughout this time.

DETAILED DESCRIPTION:
COPD is associated with disabling, progressive symptoms with episodes of rapid worsening termed acute exacerbations (AECOPD). It poses a significant global health challenge with AECOPD often resulting in the use of unscheduled care services including hospital attendance and admission. In addition to trying to prevent AECOPD, strategies have been developed to identify clinical deterioration early prompting intervention in the community with the aim of preventing unscheduled care service utilization.

Telemonitoring refers to the use of technology to monitor patients' clinical condition in their own homes. One of the proposed benefits of telemonitoring is the early detection of clinical deterioration. At present, COPD telemonitoring relies on daily symptom reporting and monitoring of basic physiological data including heart rate and pulse oximetry. However, current strategies lack specificity resulting in difficulty identifying true exacerbations from normal day to day variation.

Cough and sputum production are reported by 60-80% of COPD patients, are increased at the time of exacerbation, and are associated with accelerated lung function decline, frequent exacerbations, and earlier mortality. It has previously been demonstrated that change in cough frequency at the time of exacerbation can be detected using a cough monitor that utilizes cough classifier software to analyse ambient sound. In the context of telemonitoring, this has the potential to facilitate the early detection of clinical change using an objective measure that does not require patient effort.

Remote monitoring of COPD patients in their own homes aims to detect clinical deterioration early prompting intervention in the community with the aim of preventing utilization of unscheduled care services. Current systems do not succeed in reaching this target . A pilot study of remote cough monitoring has demonstrated that cough frequency was significantly increased during COPD exacerbation and trends in cough frequency can be detected using remote microphones and automated cough counting software. In a follow-up study, a cough-based alert system has been constructed showing promising performance. This prospective evaluation will validate the constructed system in a further COPD patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* • Clinical diagnosis of COPD using GOLD criteria.

  * 2 or more moderate and/or severe exacerbations of COPD in the previous year*.
  * Clinical stability (i.e. absence of exacerbation requiring oral corticosteroids and/or antibiotics) for at least 4 weeks prior to enrollment.
  * Current or ex-smoker with ≥10 pack-year smoking history
  * Provision of informed consent

Exclusion Criteria:

* • Children < age of 18

  * Failure to provide consent
  * Other significant comorbid medical or psychological condition that is deemed by the principal investigator to affect cough frequency or the subject's ability to comply with monitoring procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with current diagnosis of COPD who have had at least 2 moderate exacerbations of their COPD within the last year
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Acute exacerbation of COPD alert system performance | 90-190 days
  the ratio of successful alerts of acute exacerbations of COPD to false positive alerts.

SECONDARY OUTCOMES:
number of successfull alerts of Acute exacerbations of COPD | 90-180 days
  Total number of alerts of acute exacerbations of COPD identified by change in cough
Number of False positive alerts of Acute Exacerbation of COPD | 90-180 days
  Total number of Acute exacerbation alerts detected by monitoring cough that didn't result in a acute exacerbation of COPD
correlation cough counts with questionnaire data | 90-180 days
  correlate Hull airway reflux questionnaire scores, cough visual analgue scale with average cough counts

CONTACTS AND LOCATIONS:
Locations (1):
- Redspiratory mMedicine, First Floor, Daisy Building, Castle Hill Hospital, Cottingham, East Yorkshiure, United Kingdom

REFERENCES:
- [Result] Kessler R, Partridge MR, Miravitlles M, Cazzola M, Vogelmeier C, Leynaud D, Ostinelli J. Symptom variability in patients with severe COPD: a pan-European cross-sectional study. Eur Respir J. 2011 Feb;37(2):264-72. doi: 10.1183/09031936.00051110. Epub 2010 Nov 29. PMID 21115606
- [Result] de Oliveira JC, de Carvalho Aguiar I, de Oliveira Beloto AC, Santos IR, Filho FS, Sampaio LM, Donner CF, Oliveira LV. Clinical significance in COPD patients followed in a real practice. Multidiscip Respir Med. 2013 Jun 28;8(1):43. doi: 10.1186/2049-6958-8-43. PMID 23806051
- [Result] Burgel PR, Nesme-Meyer P, Chanez P, Caillaud D, Carre P, Perez T, Roche N; Initiatives Bronchopneumopathie Chronique Obstructive (BPCO) Scientific Committee. Cough and sputum production are associated with frequent exacerbations and hospitalizations in COPD subjects. Chest. 2009 Apr;135(4):975-982. doi: 10.1378/chest.08-2062. Epub 2008 Nov 18. PMID 19017866
- [Result] Vestbo J, Prescott E, Lange P. Association of chronic mucus hypersecretion with FEV1 decline and chronic obstructive pulmonary disease morbidity. Copenhagen City Heart Study Group. Am J Respir Crit Care Med. 1996 May;153(5):1530-5. doi: 10.1164/ajrccm.153.5.8630597.
- [Result] Ekberg-Aronsson M, Pehrsson K, Nilsson JA, Nilsson PM, Lofdahl CG. Mortality in GOLD stages of COPD and its dependence on symptoms of chronic bronchitis. Respir Res. 2005 Aug 25;6(1):98. doi: 10.1186/1465-9921-6-98. PMID 16120227